CLINICAL TRIAL: NCT01113021
Title: Phase 1. Muscle Genic Expression Under Strength Training and Photostimulated by Laser.
Brief Title: Study of Effects of Low Level Laser Therapy in the Physical Training and the Muscle Responses in Humans.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Universidade Federal de Sao Carlos (Other)
Other Study IDs: CAAE 0072.0.135.000-08
Record Dates: First submitted 2010-04-28; First posted 2010-04-29 (Estimated); Last update posted 2010-04-29 (Estimated); Status verified 2008-08

CONDITIONS: Healthy Young Male Volunteers; Non Athletes; Free of Metabolic Disease; Joint, Bone and Muscles of Lower Limbs Free of Any Disease

ARMS (1):
- LLLT and Physical Strength training in Humans (Experimental)
  Interventions: Device: Photon stimulation by low level laser therapy

INTERVENTIONS:
Device: Photon stimulation by low level laser therapy

SUMMARY:
The hypothesis of this study is that a chronic program of physical strength

training, associates to effects of low level laser therapy (LLLT) can,

possibly, provide changes in genic expression of muscle and to promote an

enhancement of anaerobic muscle performance in humans.

ELIGIBILITY:
Inclusion Criteria:

* healthy young male volunteers;
* non-athletic physical activity;
* Body Mass Index (BMI) under 26;
* no prescription medicine or dietary supplement use (such as muscle mass builders.

Exclusion Criteria:

* metabolic disease;
* joint, bone and muscles of lower limbs with any disease

Ages: 18 Years to 28 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of São Carlos, São Carlos, São Paulo, Brazil

REFERENCES:
- [Background] Leal Junior EC, Lopes-Martins RA, Dalan F, Ferrari M, Sbabo FM, Generosi RA, Baroni BM, Penna SC, Iversen VV, Bjordal JM. Effect of 655-nm low-level laser therapy on exercise-induced skeletal muscle fatigue in humans. Photomed Laser Surg. 2008 Oct;26(5):419-24. doi: 10.1089/pho.2007.2160. PMID 18817474
- [Background] Leal Junior EC, Lopes-Martins RA, Vanin AA, Baroni BM, Grosselli D, De Marchi T, Iversen VV, Bjordal JM. Effect of 830 nm low-level laser therapy in exercise-induced skeletal muscle fatigue in humans. Lasers Med Sci. 2009 May;24(3):425-31. doi: 10.1007/s10103-008-0592-9. Epub 2008 Jul 23. PMID 18649044
- [Background] Leal Junior EC, Lopes-Martins RA, Baroni BM, De Marchi T, Taufer D, Manfro DS, Rech M, Danna V, Grosselli D, Generosi RA, Marcos RL, Ramos L, Bjordal JM. Effect of 830 nm low-level laser therapy applied before high-intensity exercises on skeletal muscle recovery in athletes. Lasers Med Sci. 2009 Nov;24(6):857-63. doi: 10.1007/s10103-008-0633-4. Epub 2008 Dec 5. PMID 19057981
- [Background] Leal Junior EC, Lopes-Martins RA, Baroni BM, De Marchi T, Rossi RP, Grosselli D, Generosi RA, de Godoi V, Basso M, Mancalossi JL, Bjordal JM. Comparison between single-diode low-level laser therapy (LLLT) and LED multi-diode (cluster) therapy (LEDT) applications before high-intensity exercise. Photomed Laser Surg. 2009 Aug;27(4):617-23. doi: 10.1089/pho.2008.2350. PMID 19302015
- See also: Related Info — http://ufscar.br
- See also: Related Info — http://cnpq.br
- See also: Related Info — http://fapesp.br